CLINICAL TRIAL: NCT00604760
Title: A Phase 2a, Multi-Center, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety and Efficacy of MEM 3454 as Adjunctive Treatment in Combination With a Preexisting Antipsychotic in Patients With Cognitive Impairment Associated With Schizophrenia
Brief Title: Study to Evaluate the Safety and Efficacy of MEM 3454 as Adjunctive Treatment in Combination With a Preexisting Antipsychotic in Patients With Cognitive Impairment Associated With Schizophrenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Memory Pharmaceuticals (Industry)
Responsible Party: Amy S. Domanowski, Ph.D., Head Regulatory Affairs, Memory Pharmaceuticals Corp.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEM 3454-101
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Cognitive Impairment Associated With Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental)
  Interventions: Drug: MEM 3454
- B (Experimental)
  Interventions: Drug: MEM 3454
- C (Experimental)
  Interventions: Drug: MEM 3454
- D (Placebo Comparator)
  Interventions: Drug: Placebo for MEM 3454

INTERVENTIONS:
Drug: MEM 3454 — Capsule 5 mg once a day
  Arms: A
Drug: MEM 3454 — Capsule 15 mg once a day
  Arms: B
Drug: MEM 3454 — Capsule 50 mg once a day
  Arms: C
Drug: Placebo for MEM 3454 — Capsule once a day
  Arms: D

SUMMARY:
To establish the proof of concept that MEM 3454, used as add-on pharmacotherapy, is a safe and effective treatment in patients with cognitive impairment associated with schizophrenia (CIAS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (any subtype), assessed using a structured interview.
* At least one month on the same dose of antipsychotic medication.
* Clinically stable, as judged by the investigator, and in a non-acute phase for at least 12 weeks.
* Able to provide informed consent.
* Fluent in English.
* Smokers and non-smokers.

Exclusion Criteria:

* First 3 years of schizophrenia diagnosis.
* Current risk of suicide, or history of suicidal behavior within the last 6 months.
* Hospitalized for psychiatric symptoms in the past 3 months.
* Other psychiatric diagnoses.
* Substance abuse/dependence (other than nicotine or caffeine) within the last 6 months according.
* Nicotine replacement therapy, smoking cessation medications or remedies, including Varenicline (Chantix).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the total composite score of the MATRICS cognitive battery at week 8. | Change from baseline at wk 8.

SECONDARY OUTCOMES:
Change from baseline in the total composite score of the MATRICS cognitive battery at Weeks 4 and 10 | Change from baseline - weeks 4 and 10
Change from baseline on the various cognition tests at Weeks 4, 8 and 10 | Change from baseline at Weeks 4, 8 and 10
Functional Assessments Change from baseline on the following tests at Week 8 and 10: UPSA-2 and PSP | Change from baseline at weeks 8 and 10
Adverse events | weeks 2, 4, 6, 8, 10

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Telecare-Cresta Loma, Lemon Grove, California
  - Newport Bay Hospital, Newport Beach, California
  - Excell Research, Oceanside, California
  - Pasadena Research Institute, Pasadena, California
  - BHC Alhambra Hospital, Rosemead, California
  - California Clinical Trials Medical Group, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Coastal Communities Hospital, Santa Ana, California
  - Collaborative NeuroScience Network, Inc., Torrance, California
  - Aventura Hospital, Aventura, Florida
  - Fort Lauderdale Hospital, Fort Lauderdale, Florida
  - Aventura Hospital, Miami, Florida
  - TuKoi Clinical Research, Miami, Florida
  - Professional Clinical Research, Inc. c/o Segal Institute for Clinical Research, North Miami, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Berwyn Rehabilitation Center, Berwyn, Illinois
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Chinmay K. Patel, DO, Hoffman Estates, Illinois
  - American Medical Research, Inc., Oak Brook, Illinois
  - Clinical Research Institute, Wichita, Kansas
  - Parkwood Behavioral Health System, Olive Branch, Mississippi
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - CRI Worldwide, LLC at Lourdes Medical Center of Burlington County, Willingboro, New Jersey
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Arthur P. Noyes Research Foundation, Norristown, Pennsylvania
  - CRC Worldwide, LLC, Philadelphia, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Centerstone, Madison, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Vogelfanger and Struble Clinic, Memphis, Tennessee
  - Lakeside Behavioral Health System, Memphis, Tennessee
  - Centerstone - Ella Hayes Center, Nashville, Tennessee
  - Vanderbilt Psychiatric Hospital, Nashville, Tennessee
  - Centerstone - Frank Luton Center, Nashville, Tennessee
  - Texas NeuroRehab Center, Pecos Unit, Austin, Texas
  - Community Clinical Reserarch, Inc., Austin, Texas
  - FutureSearch Trials, Austin, Texas
  - University Hills Clinical Research, Irving, Texas
  - Poplar Springs Hospital, Petersburg, Virginia
  - International Clinical Research Associates, LLC, Richmond, Virginia
  - Pacific Institute of Medical Sciences, Bothell, Washington

REFERENCES:
- [Background] Buchanan RW, Davis M, Goff D, Green MF, Keefe RS, Leon AC, Nuechterlein KH, Laughren T, Levin R, Stover E, Fenton W, Marder SR. A summary of the FDA-NIMH-MATRICS workshop on clinical trial design for neurocognitive drugs for schizophrenia. Schizophr Bull. 2005 Jan;31(1):5-19. doi: 10.1093/schbul/sbi020. Epub 2005 Feb 16. PMID 15888422
- [Background] Olincy A, Harris JG, Johnson LL, Pender V, Kongs S, Allensworth D, Ellis J, Zerbe GO, Leonard S, Stevens KE, Stevens JO, Martin L, Adler LE, Soti F, Kem WR, Freedman R. Proof-of-concept trial of an alpha7 nicotinic agonist in schizophrenia. Arch Gen Psychiatry. 2006 Jun;63(6):630-8. doi: 10.1001/archpsyc.63.6.630. PMID 16754836
- See also: MATRICS Tests — http://www.matricsinc.org/